CLINICAL TRIAL: NCT02398526
Title: PARABO - Pain Evaluation in Radium-223 (Xofigo®) Treated mCRPC Patients With Bone Metastases - a Non-interventional Study in Nuclear Medicine Centers
Brief Title: Pain Evaluation in Radium-223 Treated Castration Resistant Prostate Cancer Patients With Bone Metastases
Acronym: PARABO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17550; XF1412DE (Other: Company internal)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Castration-Resistant Prostatic Cancer
Keywords: Observational study; Bone metastases; Hormone Refractory Prostatic Cancer; Xofigo; Radium-223
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223 dichloride: Male patients with a diagnosis of CRPC with symptomatic bone metastases without known visceral metastases will be enrolled after the decision for treatment with Radium-223 has been made by the attending physician according to his/her medical practice.
  Interventions: Drug: Radium-223 dichloride, (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride, (Xofigo, BAY88-8223) — Dosage and treatment duration according to the decision of the treating physician

SUMMARY:
This observational prospective single arm cohort study is designed to assess pain and bone pain related quality of life of metastatic Castration Resistant Prostate Cancer (mCRPC) patients receiving Radium-223 in a real life nuclear medicine practice setting. In addition, overall survival, time to next tumor treatment (TTNT), time to first symptomatic skeletal event (SSE), course of blood counts, and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients diagnosed with CRPC with symptomatic bone metastases without known visceral metastases
* Decision to initiate treatment with Radium-223 was made as per investigator's routine treatment practice

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice or participating in another observational study with Xofigo

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of castration resistant prostate cancer patients with bone metastases treated with Radium-223.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Pain response | Up to 6 months
  Determined by the worst pain item on the Brief Pain Inventory - Short Form (BPI-SF) patient questionnaire. A clinically meaningful pain response is defined as an improvement of two points from the baseline BPI-SF worst pain score at any post-baseline assessment.

SECONDARY OUTCOMES:
Change of pain over time | Up to 6 months from baseline
  Determined by evaluating the worst pain item as well as the subscale scores for pain severity and pain interference as determined by patient responses on the BPI-SF questionnaire.
Change in bone pain related quality of life | Up to 6 months from baseline
  As determined by patient responses on the bone pain specific Functional Assessment of Cancer Therapy Quality of Life Measurement in patients with bone pain (FACT-BP) questionnaire
Pain control rate | Up to 6 months
  As determined by the worst pain item on the BPI-SF patient questionnaire. Pain control is defined as no increase by two points from the baseline BPI-SF worst pain score.
Pain progression rate | Up to 6 months
  As determined by the worst pain item on the BPI-SF patient questionnaire. Pain progression is defined as an increase by two points from the baseline BPI-SF worst pain score at any post baseline assessment.
Time to first pain progression | Up to 6 months
  Defined as the time between the first injection of Radium-223 until an increase in the BPI-SF worst pain item by at least two points
Time to first opioid use | Up to 5.5 years
Summary description of covariates on pain response | Up to 6 months
  The following covariates will be analyzed: opioid use, assessment of extent of bone metastases, location of bone metastases,level of alkaline phosphatase at baseline, PSA (Prostate Specific Antigen) level at baseline, WHO pain score at baseline, pretreatment with chemotherapy (yes/no), pretreatment with deep androgen ablation by treatment with abiraterone or enzalutamide (yes/no), extent of bone uptake in known lesions, BSI
Relation between bone uptake in known lesions and pain palliation | Up to 6 months
  Only in patients with bone scan prior to start of treatment and a second scan during or within 6 weeks after end of Radium-223 treatment
Dosage of Radium-223 | Up to 5 months
Number of injections of Radium-223 | Up to 5 months
Course of blood count presented as percentage of patients below limit for further injections according to the local product information | Up to 5 months
Number of participants with Treatment-emergent Adverse Events (TEAE) | Up to 6 months
Time to next tumor treatment(s) (TTNT) | Up to 5.5 years
  Defined as the time from the first application of Radium-223 until start of next mCRPC treatment including e.g. chemotherapy and/or hormonal treatment
Time to first symptomatic skeletal event (SSE) | Up to 5.5 years
  Defined as the time between the first injection of Radium-223 until the occurrence of first SSE defined as the first use of external beam radiation therapy to relieve skeletal symptoms, new symptomatic pathological vertebral or non-vertebral bone fractures, spinal cord compression, or tumor-related orthopedic surgical intervention
Overall survival | Up to 5.5 years
  Defined as the time interval from the start of Radium-223 therapy to death, due to any cause. Patients alive at the end of the study will be censored at the last date known to be alive.
Bone Scan Index (BSI) as Imaging Biomarker in metastatic castration-resistant prostate cancer (mCRPC) | Up to 6 months
  Evaluated by comparing BSI values before and after Radium-223 treatment as well as by investigating the association of BSI with other outcome parameters like OS
Effect of concomitant drug treatment on pain, quality of life, and overall survival | Up to 5.5 years
  Exploration of the influence of abiraterone, enzalutamide, opioids and denosumab on OS by number of injections (5-6 vs. 1-4)
Time from castration resistance to treatment with Radium-223 | First treatment
  Time from verified castration resistance to first injection of Radium-223
Description of covariates on duration of therapy | Up to 6 months
  Description of covariates on duration of therapy (to get ≥ 5 injections versus ≤ 4 injections) of mCRPC patients during treatment with Radium-223.
Factors positively influencing mCRPC patients to get ≥ 5 injections versus ≤ 4 injections | Up to 6 months
  (e.g. concomitant use of antihormonal therapy, no pre-treatment of chemotherapy)
Incidence of pathological fractures, non-pathological fractures and bone associated events during treatment and follow up | Up to 5.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany

REFERENCES:
- [Derived] Palmedo H, Ahmadzadehfar H, Eschmann S, Niesen A, Schonberger J, Barsegian V, Liepe K, Mottaghy FM, Guan R, Pinkert J, Sandstrom P, Herrmann K. Pain Outcomes in Patients with Metastatic Castration-Resistant Prostate Cancer Treated with 223Ra: PARABO, a Prospective, Noninterventional Study. J Nucl Med. 2023 Sep;64(9):1392-1398. doi: 10.2967/jnumed.123.265557. Epub 2023 Jun 29. PMID 37385670
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/